CLINICAL TRIAL: NCT00489697
Title: Medical and Economical Evaluation of Contrast-enhanced Ultrasound Imaging for the Early Estimate of Bevacizumab Effect on Colorectal Cancer Liver Metastases
Brief Title: Evaluation of Contrast-enhanced Ultrasound Imaging for the Early Estimate of Bevacizumab Effect on Colorectal Cancer Liver Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Directrice de la Recherche et des Affaires Médicales, University Hospital Tours
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INCA06-FT/STIC-AVASTIN
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; hepatic metastases; bevacizumab; anti-angiogenic agent; chemotherapy regimens; tumor vascularity; Contrast-enhanced ultrasound
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (single arm) (Experimental): patient with histologically confirmed colorectal tumor treated in first line by a bevacizumab based chemotherapy
  Interventions: Device: real-time contrast-enhanced ultrasound imaging (CEUS)

INTERVENTIONS:
Device: real-time contrast-enhanced ultrasound imaging (CEUS) — Real time contrast enhanced sonography was performed using an ultrasound dedicated system after bolus injection of 1.2 and 2x2.4 ml Sonovue ® (Bracco, Milan, Italy)

SUMMARY:
Bevacizumab, an anti-angiogenic agent, plus fluorouracil based chemotherapy is considered a new standard for the treatment of metastatic colorectal cancer. Contrast-enhanced ultrasound with gas-encapsulated microbubbles can be used to assess tumour vascularity, particularly hepatic metastases, and may become a useful tool for monitoring anti-angiogenic therapies. The aim of this prospective, multicenter, non-randomized study is to evaluate the usefulness of hepatic contrast-enhanced ultrasound to predict response to bevacizumab based chemotherapy in patient with metastatic colorectal cancer. The primary objective of this study is to compare the functional vascular changes related to bevacizumab based chemotherapy and evaluated by hepatic contrast-enhanced ultrasound with classic RECIST criteria. The secondary objectives are to do a characterization of the pharmacokinetic of bevacizumab, to explore the pharmacodynamic effects of bevacizumab on functional vascular changes of hepatic metastases evaluated by hepatic contrast-enhanced ultrasound and to analyze the possible relationships between treatment efficacy or toxicity and constitutional gene polymorphisms linked to the bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal tumor
* first line treatment by a bevacizumab based chemotherapy
* Target hepatic metastases of size lower than 5 cm and higher than 5 mm detected by conventional ultrasonography and CT or MRI
* Life expectancy > 2 months
* OMS status =< 2
* Major surgery, open biopsy, or significant traumatic injury within 28 days prior to Day 0
* informed consent signed

Exclusion Criteria:

* no target hepatic lesion detected by conventional ultrasonography
* Prior bevacizumab treatment
* Prior chemotherapy treatment for advanced disease
* Clinically significant cardiac disease (e.g. myocardial infarction or stroke within 12 months, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure not well controlled with medication, endocarditis and prosthetic valve) and any contraindications in sulphur hexafluoride administration
* Blood pressure >= 180/110 mmHg
* Daily and chronic treatment by aspirin or AINS
* Anticipation of need for major surgical procedure within 7 days prior day 0
* Urine protein > 1g/24 Hours
* Any contraindication in enhancing bevacizumab treatment
* Serious, uncontrolled, concurrent infection(s) or illness(es)
* pregnant and lactating woman

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
functional vascular changes in tumour vascularity of hepatic metastases | 2 months
Pharmacokinetic of bevacizumab between each cure of bevacizumab based chemotherapy | 2 months
ratio cost/benefit of a strategy of therapeutic monitoring by contrast-enhanced ultrasound | 2 months
evaluation of the response to bevacizumab based chemotherapy by RECIST criteria | 2 months

SECONDARY OUTCOMES:
bevacizumab-related toxicity | 2 months
response duration | 2 years
time to disease progression | 2 years
survival time | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: François TRANQUART, Professor, Principal Investigator — Centre Hospitalier de Tours, France; Thierry LECOMTE, Doctor, Principal Investigator — Centre Hospitalier de Tours, France; Bruno GIRAUDEAU, Doctor, Study Chair — INSERM CIC 2002, Centre Hospitalier de Tours, France; Emmanuel RUSCH, Professor, Study Chair — Centre Hospitalier de Tours, France
Locations (12):
- France (12):
  - CHRU d'ANGERS, Angers
  - CRLCC, Centre Paul Papin, Angers
  - CHRU Besancon, Besançon
  - Hôpital Saint-André, CHRU Bordeaux, Bordeaux
  - CRLCC, Centre René Gauducheau, Nantes Saint Herblain
  - Hôpital Pitié Salpétrière, Assistance Publique Hôpitaux de Paris, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Hôpital La Milétrie, CHRU Poitiers, Poitiers
  - Hôpital Robert Debré, CHRU Reims, Reims
  - CHU Pontchaillou, Rennes
  - CRLCC, Centre Eugène Marquis, Rennes
  - Chru Tours, Tours

REFERENCES:
- [Background] Bleuzen A, Huang C, Olar M, Tchuenbou J, Tranquart F. Diagnostic accuracy of contrast-enhanced ultrasound in focal lesions of the liver using cadence contrast pulse sequencing. Ultraschall Med. 2006 Feb;27(1):40-8. doi: 10.1055/s-2005-858944. PMID 16470478
- [Background] Forsberg F, Ro RJ, Potoczek M, Liu JB, Merritt CR, James KM, Dicker AP, Nazarian LN. Assessment of angiogenesis: implications for ultrasound imaging. Ultrasonics. 2004 Apr;42(1-9):325-30. doi: 10.1016/j.ultras.2003.12.026. PMID 15047306
- [Background] Broillet A, Hantson J, Ruegg C, Messager T, Schneider M. Assessment of microvascular perfusion changes in a rat breast tumor model using SonoVue to monitor the effects of different anti-angiogenic therapies. Acad Radiol. 2005 May;12 Suppl 1:S28-33. doi: 10.1016/j.acra.2005.02.021. No abstract available. PMID 16106543
- [Background] Niermann KJ, Fleischer AC, Donnelly EF, Schueneman AJ, Geng L, Hallahan DE. Sonographic depiction of changes of tumor vascularity in response to various therapies. Ultrasound Q. 2005 Jun;21(2):61-7; quiz 149, 153-4. PMID 15905816
- [Background] Preda A, Novikov V, Moglich M, Turetschek K, Shames DM, Brasch RC, Cavagna FM, Roberts TP. MRI monitoring of Avastin antiangiogenesis therapy using B22956/1, a new blood pool contrast agent, in an experimental model of human cancer. J Magn Reson Imaging. 2004 Nov;20(5):865-73. doi: 10.1002/jmri.20184. PMID 15503324
- [Background] Gerber HP, Ferrara N. Pharmacology and pharmacodynamics of bevacizumab as monotherapy or in combination with cytotoxic therapy in preclinical studies. Cancer Res. 2005 Feb 1;65(3):671-80. PMID 15705858
- [Background] Zondor SD, Medina PJ. Bevacizumab: an angiogenesis inhibitor with efficacy in colorectal and other malignancies. Ann Pharmacother. 2004 Jul-Aug;38(7-8):1258-64. doi: 10.1345/aph.1D470. Epub 2004 Jun 8. PMID 15187215
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Derived] Mazard T, Mollevi C, Loyer EM, Leger J, Chautard R, Bouche O, Borg C, Armand-Dujardin P, Bleuzen A, Assenat E, Lecomte T. Prognostic value of the tumor-to-liver density ratio in patients with metastatic colorectal cancer treated with bevacizumab-based chemotherapy. A post-hoc study of the STIC-AVASTIN trial. Cancer Imaging. 2024 Jun 17;24(1):77. doi: 10.1186/s40644-024-00722-7. PMID 38886836
- [Derived] Lobet S, Caulet M, Paintaud G, Azzopardi N, Desvignes C, Chautard R, Borg C, Capitain O, Ferru A, Bouche O, Lecomte T, Ternant D. Confounding mitigation for the exposure-response relationship of bevacizumab in colorectal cancer patients. Br J Clin Pharmacol. 2024 Apr;90(4):976-986. doi: 10.1111/bcp.15983. Epub 2023 Dec 29. PMID 38072829
- [Derived] Jary M, Lecomte T, Bouche O, Kim S, Dobi E, Queiroz L, Ghiringhelli F, Etienne H, Leger J, Godet Y, Balland J, Lakkis Z, Adotevi O, Bonnetain F, Borg C, Vernerey D. Prognostic value of baseline seric Syndecan-1 in initially unresectable metastatic colorectal cancer patients: a simple biological score. Int J Cancer. 2016 Nov 15;139(10):2325-35. doi: 10.1002/ijc.30367. Epub 2016 Aug 13. PMID 27472156